CLINICAL TRIAL: NCT02828553
Title: CHF Inpatient Ambulation Trial
Status: Completed | Type: Observational
Sponsor: Lancaster General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CHF Inpatient Ambulation Trial
Record Dates: First submitted 2016-06-07; First posted 2016-07-11 (Estimated); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Heart Failure
Keywords: Wearable device; Fitbit; Inpatient
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control Group - Usual Care: At the start of the study, subjects will be enrolled in usual care when admitted to the heart failure unit following standard protocols.
- Intervention Group - Aggressive Ambulation: After a washout period and transition to a new aggressive ambulation protocol, subjects will be enrolled to usual care + aggressive planned ambulation with a trained mobility aide.
  Interventions: Other: Aggressive planned ambulation with a mobility aide

INTERVENTIONS:
Other: Aggressive planned ambulation with a mobility aide — A trained mobility aide will provide aggressive ambulation at least 3X per day for all patients on the heart failure unit
  Groups: Intervention Group - Aggressive Ambulation

SUMMARY:
There is an overwhelming amount of deconditioning that occurs during the hospitalization to a patient admitted with a primary diagnosis of congestive heart failure. The goals of this study are to determine if monitored activity and aggressive mobility provides improved outcomes in hospitalized heart failure patients.

DETAILED DESCRIPTION:
By implementing an ambulatory study, the goal is to decrease the hospital length of stay by half of a day, decrease the percentage of patients being discharged to an extended nursing care facility, and improve quality of life for the patient. Fiscal year 2014 the average length of stay for a CHF patient at Lancaster General Health was 6.0, and as of fiscal year 2015 this was decreased to 5.8. According to Harlan M Krumbholz's theory of post hospital syndrome, patients are subjected to a time of increased risk of impaired stamina, coordination, strength and readmission for about thirty days after discharge due to deconditioning during their hospitalization. By implementing the ambulatory study, the hope is to prevent such extensive deconditioning to help improve the patient's quality of life after discharge; thereby reducing length of stay, discharges to skilled nursing facilities, 30 day readmissions and costs.

The advent of wearable activity and/or health monitors in the health and fitness industry segment has the potential to revolutionize the industry. More importantly, these devices allow new variables to be collected to provide an impact on patients' care and outcome such as steps taken per day.

The intention of the ambulation study is to prevent hospital acquired deconditioning; which in turn would not only decrease the length of stay, but also improve the discharge disposition and place them at home rather than hospice, an extended care facility or rehab. Not only is the intent of the study to decrease the length of stay and also improve the patient's disposition, but also improve their quality of life. In addition, the study will test the effectiveness of the addition of a mobility aide to assist with patients walking on the nursing units.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of heart failure
* The heart group as attending or consultant
* Patient on 5 West at the time of admission
* Admission diagnosis of heart failure
* Age ≥ 18
* Initial assessment completed within 10 hours of admission by a registered nurse

Exclusion Criteria:

* Patient admitted from acute rehabilitation or skilled nursing facility
* Altered weight bearing or unable to complete initial 2 minute walk test
* Unwilling or unable to participate or consent
* Acute delirium or dementia by history
* Hospice or actively dying
* Ventricular assist device or listed for heart transplantation
* Inotrope dependence
* Active ischemia
* Heart rate (HR) <50 or >130 at rest
* Blood pressure (BP) <80 or >180 at rest
* Pulse oximetry <88% at rest
* Patient is in isolation for multi-drug resistant organism such as MRSA or C-diff

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients entering the Lancaster General Hospital heart failure unit (5 East or 5 West) will be evaluated with a 2 minute walk test and if able to complete this test will be offered the opportunity to enroll/consent for participation.
Sampling Method: Non-Probability Sample
Enrollment: 352 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Walk distance | Through study completion, an average of 5 days
  Walk distance using a 2-minute walk test will be assessed at admission and again at discharge. A clear starting and stopping point will be made with distance marked every 10 feet. A chair with armrests will be at the starting and stopping point of the walk distance. The designated area will be between 5 East and 5 West which will be standard for each patient. After the assessment the nurse will document the total patient's distance to the nearest 10 feet. Example "Ms. Smith walked 100 feet with 3 stops in 2 minutes." The patient will have a repeat 2 minute walk test on the day of discharge using the same criteria. For the walk test:
  * Gait belt must be used
  * Patient will be allowed to stop, lean on the wall and rest, but if requires sitting, terminates the 2 minute walk distance.
  * IV medications on hold is able
Steps per day | Through study completion, an average of 5 days
  Steps per day for each day in the hospital will be measured in 15-minute intervals from admission to discharge using a Fitbit device (wearable device on the wrist). Data will be downloaded from the Fitbit upon discharge.

SECONDARY OUTCOMES:
Disposition at Discharge | At discharge/completion of study; an average of 5 days after admission
  Discharge disposition to home, skilled care/nursing care, etc. will be tracked.
Readmission within 30 days | 30 Days after discharge
  Readmission within 30 days of discharge
Falls | Through study completion, an average of 5 days
  Record any falls or near falls for subjects enrolled in the study during hospital stay from admission to discharge
Length of Stay | Through study completion, an average of 5 days
  Calculation of length of stay from hour/day of admission to hour/day of discharge

CONTACTS AND LOCATIONS:
Overall Officials: Justin Roberts, DO, Principal Investigator — Lancaster General Hospital; Lisa Rathman, CRNP, Principal Investigator — Lancaster General Hospital; Dana Irwin, BSN, RN, Principal Investigator — Lancaster General Hospital; Michael Killinger, MSN, RN, Principal Investigator — Lancaster General Hospital; Nathaniel Baker, DPT, Principal Investigator — Lancaster General Hospital; Michael Horst, PhD, Principal Investigator — Lancaster General Hospital
Locations (1):
- Lancaster General Hospital, Lancaster, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Study results will be published in aggregate.